CLINICAL TRIAL: NCT01393496
Title: Effects of Transfusion Thresholds on Neurocognitive Outcome of Extremely Low Birth Weight Infants (ETTNO)- a Blinded Randomized Controlled Multicenter Trial
Brief Title: Effects of Transfusion Thresholds on Neurocognitive Outcome of Extremely Low Birth Weight Infants
Acronym: ETTNO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Axel Franz, Coordinating Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFG Fr 1455/6-1; 2010-021576-28 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Anemia of Prematurity
Keywords: prematurity; anemia; transfusion
MeSH Terms: conditions — Anemia; Premature Birth | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "liberal" transfusion triggers (Experimental): "liberal" guidelines for red blood cell transfusions
  Interventions: Other: red blood cell transfusion
- "restrictive" transfusion triggers (Active Comparator): "restrictive" guidelines for red blood cell transfusions
  Interventions: Other: red blood cell transfusion

INTERVENTIONS:
Other: red blood cell transfusion — Implementation of "liberal" guidelines for red blood cell transfusions in extremely low birth weight infants
  Arms: "liberal" transfusion triggers
Other: red blood cell transfusion — Implementation of "restrictive" guidelines for red blood cell transfusions in extremely low birth weight infants
  Arms: "restrictive" transfusion triggers

SUMMARY:
To compare the effect of restrictive versus liberal red blood cell transfusion thresholds on long-term neurodevelopmental outcome in extremely low birth weight infants.

DETAILED DESCRIPTION:
Extremely low birth weight (ELBW) infants uniformly develop anemia of prematurity and frequently require multiple red blood cell transfusions (RBCT) during neonatal intensive care. The criteria currently applied to indicate RBCT in this population are based on expert opinion rather than evidence and conclusive data of long-term effects of RBCT practices do not exist. Both, giving RBCT to improve oxygen carrying capacity and restricting RBCT to avoid RBCT associated risks and costs potentially impair long-term development. The proposed blinded randomized controlled trial was designed and will be powered to compare the effect of restrictive versus liberal red blood cell transfusion guidelines on long-term neurodevelopmental outcome in ELBW infants. ELBW infants will be randomized to receive RBCT according to liberal or restrictive RBCT guidelines, which both reflect current practice in Germany and aim for a clinically relevant difference in mean hemoglobin concentrations. The primary outcome measure is the incidence of death or major neurodevelopmental impairment determined at 24 months of age corrected for prematurity. Key secondary outcomes are the incidences of individual components of the composite primary outcome, the mental and physical developmental index scores of the Bayley Scales of Infant Development (II edition), and growth. Safety analyses will assess the incidences of all major diseases of prematurity. The results of this trial may help to improve the quality of life of these patients and reduce long-term health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight of 400 - 999g

Exclusion Criteria:

* Missing written parental consent.
* Gestational age > 29 + 6/7 weeks
* Major congenital anomalies (including chromosomal aberrations, cyanotic congenital heart defects, syndromes likely affecting long-term outcome, and major congenital malformations requiring surgical correction during newborn period).
* Infants who died before 48 hours, infants in whom the clinical decision to withhold intensive care was made, infants who were not considered viable
* Participation in another study with ongoing use of an unlicensed investigational product from 28 days before study enrollment until the end of the study

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1013 (Actual)
Dates: Start 2011-07; Primary Completion 2017-04-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of death or major neurodevelopmental impairment | 24 months of age corrected for prematurity
  The primary outcome measure of this study will be the incidence of death or major neurodevelopmental impairment determined at 24 months of age corrected for prematurity (where major neurodevelopmental impairment is defined as any of the following: cognitive delay defined as mental developmental index (MDI) score of the Bayley Scales of Infant Development (2nd edition) < 85, cerebral palsy, or severe visual or hearing impairment

CONTACTS AND LOCATIONS:
Overall Officials: Axel R Franz, MD, Principal Investigator — University Hospital of Tuebingen
Locations (32):
- Neonatalklinikken, Copenhagen, Denmark
- Germany (31):
  - University Hospital of Aachen, Aachen
  - Children's Hospital, Augsburg
  - Vivantes Children's Hospital, Berlin
  - Charité University Children's Hospital, Berlin
  - University Children's Hospital, Bochum
  - Children's Hospital, Cologne
  - University Children's Hospital, Cologne
  - Children's Hospital, Datteln
  - University Children's Hospital, Dresden
  - University of Duesseldorf, Düsseldorf
  - Helios Children's Hospital, Erfurt
  - Children's Hospital, Erlangen
  - University Children's Hospital, Essen
  - University Children's Hospital, Frankfurt
  - University Children's Hospital, Giessen
  - University of Greifswald, Greifswald
  - Children's Hospital Eppendorf, Hamburg
  - Children's Hospital Altona, Hamburg
  - Children's Hospital, Hanover
  - University Hospital of Leipzig, Leipzig
  - University of Luebeck, Lübeck
  - University Children's Hospital, Magdeburg
  - University Hospital of Marburg, Marburg
  - University Children's Hospital, Munich
  - University Children's Hospital, Münster
  - Children's Hospital, Nuremberg
  - Children's Hospital St. Hedwig, Regensburg
  - DRK Kinderklinik, Siegen
  - Children's Hospital, Stuttgart
  - University Hospital of Tuebingen, Tübingen
  - University Children's Hospital, Ulm

REFERENCES:
- [Background] ETTNO Investigators. The 'Effects of Transfusion Thresholds on Neurocognitive Outcome of Extremely Low Birth-Weight Infants (ETTNO)' Study: Background, Aims, and Study Protocol. Neonatology. 2012 Jun;101(4):301-305. doi: 10.1159/000335030. Epub 2012 Jan 27. PMID 22298226
- [Result] Franz AR, Engel C, Bassler D, Rudiger M, Thome UH, Maier RF, Krageloh-Mann I, Kron M, Essers J, Buhrer C, Rellensmann G, Rossi R, Bittrich HJ, Roll C, Hohn T, Ehrhardt H, Avenarius S, Korner HT, Stein A, Buxmann H, Vochem M, Poets CF; ETTNO Investigators. Effects of Liberal vs Restrictive Transfusion Thresholds on Survival and Neurocognitive Outcomes in Extremely Low-Birth-Weight Infants: The ETTNO Randomized Clinical Trial. JAMA. 2020 Aug 11;324(6):560-570. doi: 10.1001/jama.2020.10690. PMID 32780138
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Franz AR, Engel C, Bassler D, Rudiger M, Thome UH, Maier RF, Krageloh-Mann I, Essers J, Buhrer C, Bittrich HJ, Roll C, Hohn T, Ehrhardt H, Boettger R, Korner HT, Stein A, Neuberger P, Henriksen TB, Greisen G, Poets CF; ETTNO Investigators. Effects of liberal versus restrictive transfusion strategies on intermittent hypoxaemia in extremely low birthweight infants: secondary analyses of the ETTNO randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2025 Oct 17;110(6):564-570. doi: 10.1136/archdischild-2024-327643. PMID 40139741
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836